CLINICAL TRIAL: NCT03309878
Title: A Phase I and Randomized Phase II Study of KW-0761 (Mogamulizumab) and MK-3475 (Pembrolizumab) in Relapsed, Refractory Diffuse Large-B Cell Lymphoma
Brief Title: Mogamulizumab and Pembrolizumab in Treating Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01865; NCI-2017-01865 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-018; 10106 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10106 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2017-10-13; First posted 2017-10-16 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent Transformed B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Transformed B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — mogamulizumab; Immunoglobulin G; Disulfides; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (pembrolizumab, mogamulizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and mogamulizumab IV over 60 minutes on days 1, 8, and 15 of cycle 1, then day 1 of subsequent courses. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Mogamulizumab; Biological: Pembrolizumab
- Arm II (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Mogamulizumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(CC Chemokine Receptor CCR4) (Human-Mouse Monoclonal KW-0761 Heavy Chain), Disulfide With Human-Mouse Monoclonal KW-0761 Kappa-Chain, Dimer; KM8761; KW-0761; Mogamulizumab-kpkc; Poteligeo
  Arms: Arm I (pembrolizumab, mogamulizumab)
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Keytruda; Lambrolizumab; MK-3475; Pembrolizumab Biosimilar BCD-201; SCH 900475

SUMMARY:
This phase I/II trial studies the best dose and side effects of mogamulizumab in combination with pembrolizumab and to see how well they work in treating patients with diffuse large B cell lymphoma that have come back after a period of improvement (relapsed) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as mogamulizumab and pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of KW-0761 (mogamulizumab) when administered in combination with MK-3475 (pembrolizumab) in patients with relapsed, refractory diffuse large B-cell lymphoma. (Phase I) II. To assess the safety and tolerability of KW-0761 (mogamulizumab) when administered in combination with MK-3475 (pembrolizumab) in patients with relapsed, refractory diffuse large B-cell lymphoma. (Phase I) III. To assess the progression-free survival of KW-0761 (mogamulizumab) when administered in combination with MK-3475 (pembrolizumab) compared to MK-3475 (pembrolizumab) alone in patients with relapsed and refractory diffuse large B-cell lymphomas. (Phase II)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. (Phase I) II. To assess the overall response rate, complete response rate, partial response rate, duration of response of KW-0761 (mogamulizumab) and MK-3475 (pembrolizumab) compared to MK-3475 (pembrolizumab) alone in patients with relapsed and refractory diffuse large B-cell lymphomas. (Phase II)

EXPLORATORY OBJECTIVES:

I. To determine whether the progression-free survival of KW-0761 (mogamulizumab) and MK-3475 (pembrolizumab) when administered to patients with relapsed and refractory diffuse large B-cell lymphomas differs based on the presence or absence of mutations in B2M or CD58 or amplifications in PD-L1.

II. To determine whether the progression-free survival of KW-0761 (mogamulizumab) and MK-3475 (pembrolizumab) when administered to patients with relapsed and refractory diffuse large B-cell lymphomas differs based on changes in CD8 T-cell, natural killer (NK) cell, and FoxP3+ regulatory T cell (Treg) prevalence in response to therapy as measured by immunohistochemistry.

III. To determine whether KW-0761 (mogamulizumab) and MK-3475 (pembrolizumab) alters the prevalence of peripheral blood CCR4+/FoxP3+ regulatory T-cells as well as effector CD4 and CD8 T-cells by multi-parametric flow cytometry.

OUTLINE: This is a phase I, dose-escalation study of mogamulizumab followed by a phase II study. Patients are randomized to 1 of 2 arms.

ARM I: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and mogamulizumab IV over 60 minutes on days 1, 8, and 15 of cycle 1, then day 1 of subsequent courses. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diffuse large B-cell lymphoma; all subtypes of diffuse large B-cell lymphoma are eligible, including high-grade B-cell lymphoma and diffuse large B-cell lymphoma (DLBCL) that has transformed from a prior indolent B-cell non-Hodgkin lymphoma
* Patients must have measurable disease per 2014 Lugano Classification Criteria which is defined as at least one nodal lesion measuring > 1.5 cm in greatest diameter or at least one extranodal lesion measuring > 1.0 cm in greatest diameter
* For phase 2: patients and received at least 2 prior lines of therapy and must have previously received, refused, or been deemed ineligible for autologous stem cell transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 80%)
* Absolute neutrophil count >= 1,500/mcL (if neutropenia is related to bone marrow involvement with lymphoma, the absolute neutrophil count must be >= 1,000/mcL)
* Platelets >= 75,000/mcL (if thrombocytopenia is related to bone marrow involvement with lymphoma, the platelet count must be >= 50,000/mcL)
* Hemoglobin >= 9 g/dL (if anemia is related to bone marrow involvement with lymphoma, the hemoglobin must be >= 8 g/dL)
* Total bilirubin =< 1.5 x the institutional upper limit of normal (ULN) or < 3 x the ULN for indirect bilirubin in patients with Gilbert's disease
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal OR measured or calculated creatinine clearance if creatinine > 1.5 x ULN then creatinine clearance >= 40 mL/min/1.73 m^2 as calculated by Cockcroft and Gault equation
* Life expectancy of greater than 3 months
* The effects of MK-3475 (pembrolizumab) in combination with KW-0761 (mogamulizumab) on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and 6 months after completion of MK-3475 (pembrolizumab) in combination with KW-0761 (mogamulizumab) administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of MK-3475 (pembrolizumab) in combination with KW-0761 (mogamulizumab) administration
* Submit adequate archival tissue specimen (25+ unstained slides or 2 tissue blocks) from a biopsy performed after progression of disease on most recent therapy OR subject is willing to undergo a new core or excisional biopsy to obtain evaluable tumor tissue sample for immunohistochemical assessment and sequencing for B2M loss; repeat samples may be required if adequate tissue is not provided, however, patients may still be considered for enrollment on a case by case basis following consultation with the principal investigator (PI)
* Ability to understand and the willingness to sign a written informed consent document
* Subjects with prior history of chemotherapy-induced or radiation-induced pulmonary toxicity require confirmation of diffuse capacity of the lung for carbon monoxide (DLCO) over 60% (adjusted for hemoglobin) by a pulmonary function test prior to study enrollment

Exclusion Criteria:

* Patients who have had previous systemic anti-cancer therapy within 3 weeks of registration or those who have not recovered from adverse events due to agents administered previously

  * Note: Patients are considered enrolled on the study after protocol registration and not after signing consent
* Patients who are receiving any other concurrent investigational agents
* Patient is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment; the use of physiologic doses of corticosteroids (e.g. prednisone =< 20 mg/d) may be approved after consultation with the study PI; topical or inhaled corticosteroids are allowed
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer
* Patients with active cerebral or meningeal involvement by lymphoma should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475 (pembrolizumab) or KW-0761 (mogamulizumab)
* Subject with active autoimmune disease; subjects with vitiligo, eczema, alopecia, type I diabetes mellitus, psoriasis not requiring systemic treatment, or endocrine deficiencies (such as hypothyroidism) managed with replacement hormones, including physiologic corticosteroid replacement therapy are eligible
* Has a history or currently active (non-infectious) pneumonitis that required steroids unless prior history of chemotherapy or radiotherapy induced pneumonitis meeting the eligibility criteria
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Prior allogeneic stem cell transplant (SCT)
* Patients who are planning to receive allogeneic SCT in the near future as preliminary reports suggest added toxicity in patients undergoing allogeneic stem cell transplantation after having received mogamulizumab
* Autologous SCT =< 90 days prior to first dose of study drug
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because MK-3475 (pembrolizumab) is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MK-3475 (pembrolizumab), breastfeeding should be discontinued if the mother is treated with MK-3475 (pembrolizumab); these potential risks may also apply to KW-0761 (mogamulizumab)
* MK-3475 (pembrolizumab) and KW-0761 (mogamulizumab) may have adverse effects on a fetus in utero; furthermore, it is not known if MK-3475 (pembrolizumab) or KW-0761 (mogamulizumab) has transient adverse effects on the composition of sperm; patients are excluded from this study if pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 180 days after the last dose of trial treatment
* Patients with human immunodeficiency virus (HIV) are excluded if they have a detectable viral load, are not on a stable antiretroviral regimen, have a decreased CD4+ T-cell count (< 500), or require prophylactic antibiotics for the prevention of opportunistic infections
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection

  * Note: No testing for hepatitis B and hepatitis C is required unless mandated by local health authority
* Has a known history of active tuberculosis (TB)
* Patients with significant cardiac disease (e.g., New York Heart Association [NYHA] class III-IV congestive heart failure, unstable angina, recent myocardial infarction within the last 6 months, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2023-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erel Joffe, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (8):
- United States (8):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Joffe E, Kumar A, Tuscano JM, Moskowitz AJ, Owens C, Noy A, Palomba ML, Zelenetz AD, Ni A, Sharon E, Vardhana S. Phase I Study of Mogamulizumab in Combination with Pembrolizumab in Patients with Relapsed or Refractory Non-Hodgkin Lymphoma-A National Cancer Institute Experimental Therapeutics Clinical Trials Network (NCI-ETCTN) Trial. Cancers (Basel). 2026 Jan 16;18(2):284. doi: 10.3390/cancers18020284. PMID 41595202

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Level 1: Patients receive pembrolizumab 200 mg by infusion over 30 minutes on day 1 of each cycle and mogamulizumab 1 mg/kg by infusion over 60 minutes on days 1, 8, and 15 of the first cycle, then mogamulizumab 1.5 mg/kg by infusion on day 1 of subsequent cycles. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
- Phase I Dose Level -1: Patients receive pembrolizumab 200 mg by infusion over 30 minutes on day 1 of each cycle and mogamulizumab 0.5 mg/kg by infusion over 60 minutes on days 1, 8, and 15 of the first cycle, then mogamulizumab 1 mg/kg by infusion on day 1 of subsequent cycles. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
- Phase II Arm A: Patients receive pembrolizumab 200 mg by infusion over 30 minutes on day 1 of each cycle and mogamulizumab at dose identified in Phase I given by infusion over 60 minutes on days 1, 8, and 15 of the first cycle, then mogamulizumab at dose identified in Phase I given by infusion on day 1 of subsequent cycles. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
- Phase II Arm B: Patients receive pembrolizumab 200 mg by infusion over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1 | Phase II Arm A | Phase II Arm B
Started | 4 | 4 | 0 | 0
Completed | 1 | 2 | 0 | 0
Not Completed | 3 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Did not maintain eligibility | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No enrollments to Phase II
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1 | Phase II Arm A | Phase II Arm B | Total
Number analyzed (Participants) | 4 | 4 | 0 | 0 | 8
Age, Continuous [Median (Full Range); unit: years] | 71.5 [55 to 80] | 55.5 [50 to 77] |  |  | 64.5 [50 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 |  |  | 1
  Male | 3 | 4 |  |  | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  |  | 0
  Not Hispanic or Latino | 3 | 4 |  |  | 7
  Unknown or Not Reported | 1 | 0 |  |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 0 | 1 |  |  | 1
  White | 3 | 3 |  |  | 6
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 1 | 0 |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 |  |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) or Recommended Phase II Dose (RP2D) of Mogamulizumab in Combination With Pembrolizumab (Phase I)
Description: Will be determined by dose limiting toxicity (DLT). A standard 3+3 design will be used to find the MTD or RP2D for the combination of pembrolizumab and mogamulizumab.
Time Frame: Up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1
Number analyzed (Participants) | 2 | 1
Participants
  Dose limiting toxicity occurred | 0 | 1
  Dose limiting toxicity did not occur | 2 | 0

2. Primary Outcome: Incidence of Adverse Events (Phase I)
Description: Number of incidences of grade 3-5 adverse events at least possibly related to the study intervention will be reported. Adverse events will be graded according to Common Terminology Criteria for Adverse Events version 4.03 (Version 5.0 beginning April 1, 2018).
Time Frame: Up to 25 months
Measure: Number; unit: Related Incidences
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1
Number analyzed (Participants) | 2 | 1
Related Incidences
  Experienced Grade 3 Adverse Events | 4 | 0
  Experienced Grade 4 Adverse Events | 5 | 0
  Experienced Grade 5 Adverse Events | 0 | 1

3. Primary Outcome: Progression-free Survival (PFS) (Phase II)
Description: The Kaplan Meier method will be used to estimate the median PFS.
Time Frame: From course 1 day 1 to the first date of recurrence, progression, or death due to any cause, whichever comes first, assessed up to 12 months
Population: Study closed before conducting Phase II.
Arm/Group | Phase II Arm A | Phase II Arm B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Response Rate
Description: Will be calculated along with exact 95% confidence intervals.
Time Frame: Up to 25 months
Population: Study closed before conducting Phase II.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1 | Phase II Arm A | Phase II Arm B
Number analyzed (Participants) | 2 | 1 | 0 | 0
Participants
  Experienced Complete Response | 0 | 0 |  |
  Experienced Partial Response | 0 | 0 |  |
  Experienced Stable Disease | 0 | 0 |  |
  Experienced Disease Progression | 1 | 1 |  |
  Not evaluated | 1 | 0 |  |

5. Secondary Outcome: Complete Response Rate
Description: Will be calculated along with exact 95% confidence intervals.
Time Frame: Up to 25 months
Population: Study closed before conducting Phase II.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1 | Phase II Arm A | Phase II Arm B
Number analyzed (Participants) | 2 | 1 | 0 | 0
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Partial Response Rate
Description: Will be calculated along with exact 95% confidence intervals.
Time Frame: Up to 25 months
Population: Study closed before conducting Phase II.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1 | Phase II Arm A | Phase II Arm B
Number analyzed (Participants) | 2 | 1 | 0 | 0
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Duration of Response
Description: Will be summarized by Kaplan-Meier method in patients who achieve complete response (CR) or partial response (PR).
Time Frame: Up to 25 months
Population: Participants in Phase I (Dose Levels 1 and -1) did not experience complete response or partial response. Study closed before conducting Phase II.
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1 | Phase II Arm A | Phase II Arm B
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Biomarker Analysis
Description: Performed and summarized using descriptive statistics and graphical displays at pre and post treatment time points.
Time Frame: Up to 25 months
Population: Not collected.
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1 | Phase II Arm A | Phase II Arm B
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 25 months
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level -1
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 1 (N=2) | Phase I Dose Level -1 (N=1)
Acidosis (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0
Heart failure (Cardiac disorders) | 1 (1) | 0
Colitis (Gastrointestinal disorders) | 1 (1) | 0
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0
Infusion-related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0
Ejection fraction decreased (Investigations) | 1 (1) | 0
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0
Apical ballooning (Cardiac disorders) | 1 (1) | 0
Hypotension (Vascular disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 1 (N=2) | Phase I Dose Level -1 (N=1)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 0
Confusion (Psychiatric disorders) | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Creatinine increased (Investigations) | 1 (1) | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0
Dysarthia (Nervous system disorders) | 1 (1) | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (3) | 0
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0
Fatigue (General disorders) | 2 (2) | 0
Fever (General disorders) | 2 (3) | 0
Gait disturbance (General disorders) | 1 (1) | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Hallucinations (Psychiatric disorders) | 1 (1) | 0
Headache (Nervous system disorders) | 1 (1) | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0
High degree AV block (Cardiac disorders) | 1 (1) | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypotension (Vascular disorders) | 0 | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lightheaded (Nervous system disorders) | 0 | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 0
Nausea (Gastrointestinal disorders) | 1 (1) | 0
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0
Penile bleeding (Reproductive system and breast disorders) | 1 (1) | 0
Platelet count decreased (Investigations) | 0 | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0
Presyncope (Nervous system disorders) | 1 (1) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Right bundle branch block (Cardiac disorders) | 1 (1) | 0
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 0
Weight loss (Investigations) | 1 (2) | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
White blood cell count decreased (Investigations) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT03309878/Prot_SAP_000.pdf